CLINICAL TRIAL: NCT04808024
Title: Self Myofascial Release (SMR) and Bioelectrical Activity of Muscles
Brief Title: Myofascial Release and Muscle Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Silesia (Other)
Responsible Party: Principal Investigator, Piotr Michalik, Lecturer at Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia, Katowice, Poland, Medical University of Silesia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SMR and muscle
Record Dates: First submitted 2021-03-16; First posted 2021-03-19 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2021-03

CONDITIONS: Self Myofascial Release; Muscle Tone Abnormalities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Players of amateur football leagues (Experimental): The players of amateur football leagues who will receive SelfMyofascial Release intervention
  Interventions: Procedure: SelfMyofascial Release
- Control group (No Intervention): The players of amateur football leagues who will receive no intervention

INTERVENTIONS:
Procedure: SelfMyofascial Release — Myofascial auto-release consisted of rolling the roller on a group of knee flexors for 3.5 minutes between the sciatic tumor and the knee joint in both directions, omitting the popliteal fossa. Before and after the intervention, sEMG of the biceps and gluteal muscles will be performed.
  Arms: Players of amateur football leagues

SUMMARY:
The aim of the study is to assess the impact of SMR intervention in the hamstring muscles on the activity of the biceps and gluteus muscles.

DETAILED DESCRIPTION:
The study will cover 40 men, players of amateur football leagues, aged 18 - 40. The test will include the measurement of sEMG of the biceps and gluteal muscles during the exercise, followed by myofascial self-release (SMR). Muscle sEMG was re-measured immediately after roller therapy.

ELIGIBILITY:
Inclusion Criteria:

* signing informed consent to participate in the study
* age in the range of 18-40 years

Exclusion Criteria:

* people who had orthopedic injuries to the lower limbs and the lumbar-pelvic-iliac complex in the last year
* people who reported pain in the lower limbs and the lumbar-pelvic-iliac complex on the day of the examination
* people who underwent myofascial therapy in the last 6 weeks
* people with non-specific neuromuscular disorders

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-04-21 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
1. Surface electromyography (sEMG) examination before SMR | Before the SMR intervention
  The sEMG examination of the biceps and gluteus muscles will be performed using the MyoTrace 400 recorder by Noraxon USA Inc. with a sampling frequency of 1000 Hz, using the bipolar method, in accordance with SENIAM standards.The bioelectrical activity of the muscles will be tested during the squat.
Surface electromyography (sEMG) examination immediately after SMR | Immediately after the SMR intervention
  The change in bioelectrical activity of the biceps and gluteus muscles will be performed. The bioelectrical activity of the muscles will be tested during the squat.
Surface electromyography (sEMG) examination 5 minutes after SMR | 5 minutes after the SMR intervention
  The change in bioelectrical activity of the biceps and gluteus muscles will be performed. The bioelectrical activity of the muscles will be tested during the squat.

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Dąbrowska-Galas, Study Director — Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia in Katowice, Katowice, Poland
Locations (1):
- Department of Kinesitherapy and Special Methods, SHS in Katowice, Medical University of Silesia, Katowice, Poland, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
The datasets used and / or analyzed in the present study will be available from the respective author upon reasonable request.